CLINICAL TRIAL: NCT01817426
Title: Discontinuation of Infliximab Therapy in Patients With Crohn's Disease During Sustained Complete Remission: A Multi-center, Double Blinded, Randomized, Placebo Controlled Study
Brief Title: Discontinuation of Infliximab Therapy in Patients With Crohn's Disease During Sustained Complete Remission
Acronym: STOP IT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Principal Investigator, Forskningsenheden, Mark Ainsworth, MD, professor, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 02MA
Record Dates: First submitted 2012-08-29; First posted 2013-03-25 (Estimated); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- infliximab (Active Comparator): Patients in this arm are randomized to continue IFX therapy at an unchanged dosage and frequency.
  Interventions: Drug: Infliximab
- Placebo (Placebo Comparator): Patients in this arm are randomized to receive matching placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Infliximab
  Other Names: Remicade
  Arms: infliximab
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether infliximab can favourably and safely be discontinued in patients with Crohn's disease in sustained complete clinical, biochemical, and endoscopic remission on infliximab.

Further to examine the clinical utility of measuring levels/activity of infliximab and activity of anti-infliximab Ab in patients in sustained complete remission, in order to investigate whether pharmacoimmunological data can predict the clinical outcome and rationalize therapeutic management of these patients with respect to continuation or discontinuation of infliximab therapy. Additional, to investigate the optimal time-point, out of three, to measure this activity.

DETAILED DESCRIPTION:
Recent guidelines for the management of Crohn's disease conclude that currently available data are insufficient to make firm recommendations on when and in whom to stop TNF-α antibody (TNF-α Ab) treatment after having obtained clinical remission. Further, the term "remission" is not well uniformly defined and may incorporate one or more features such as clinical remission, as assessed by CDAI, biochemical remission, endoscopical remission etc. The recently published prospective STORI study of 115 patients with luminal Crohn's disease reported that 56% of patients with Crohn's disease who had discontinued infliximab (IFX) while in clinical remission, maintained remission one year after discontinuation of therapy. Predictors of relapse included certain clinical features as well as objective biochemical and endoscopical markers of disease activity. Consistent with these data, we have recently reported that 61% of our own patients with Crohn's disease, who discontinued IFX while in complete clinical, steroid free IFX induced remission, maintained remission after one year; and half the patients were still in remission after nearly two years (median 680 days [412-948]).

A prospective randomized study of patients with Crohn's disease is necessary to confirm and extend the limited findings above, and assess whether IFX can be safely discontinued in a selected subgroup of patients with complete clinical, biochemical, and endoscopical remission.

Methods:

Study design: Prospective, double-blinded, randomized, placebo-controlled, Danish multi-center study with estimated seven Danish participating centers. Patients and treating physicians are blinded for the type of intervention.

Study population: Patients with luminal Crohn's disease in sustained complete remission on IFX.

Study treatment: Patients are randomized to either continue IFX treatment at an unchanged dosage and frequency, or alternatively to receive matching placebo. All patients will be graded for disease activity (Crohn's Disease Activity Index (CDAI), biochemical parameters, endoscopy, and/or MRI). Following screening and inclusion patients are seen after four weeks, and then every eight weeks. Endpoints are assessed at 48 weeks.

Investigators will, as explorative analyses, examine the clinical utility of measuring IFX levels and antibodies against IFX in patients with complete remission, in order to investigate whether pharmacoimmunological data can predict the clinical outcome and rationalize therapeutic management of these patients with respect to continuation or discontinuation of IFX therapy. Additional, investigators will investigate the optimal time-point out of three to measure this activity. Patients will on the day of infusion have three blood samples drawn: one just before infusion (trough), one right after the infusion (obtained from the other arm)(peak) and one an hour after infusion (C1). Samples will be measured by common solid - and fluid phase assays for this purpose, e.g. Reporter Gene Assay (RGA).

ELIGIBILITY:
Inclusion Criteria:

* Luminal Crohn's disease defined according to standardized diagnostic criteria.
* Age ≥ 18 years.
* IFX induction treatment week 0, 2, 6 followed by maintenance therapy.
* IFX treatment length minimum 12 months. Episodic therapy with IFX pause > 12 weeks is not accepted within the last year. The treatment interval in the last three months has to be of 6-10 weeks.
* Complete remission defined as:

  * CDAI score < 150 and
  * Biochemical remission, and
  * No other signs of disease activity as evaluated by endoscopic examination or by magnetic resonance imaging (MRI).
* Stable remission, judged by the treating physician, at two consecutive treatments visits corresponding 2 scheduled IFX infusions. Thus, the first visit is during IFX maintaining therapy (screening visit). The second visit is at time of inclusion corresponding time of next scheduled IFX infusion (i.e. after ≈ 8 weeks).
* No use of oral steroids within 3 months prior to inclusion.
* Concomitant therapy with other immune suppressants, except steroids, is allowed. The dosage and frequency must have been stable three months prior to inclusion and must remain stable throughout the study period.

Exclusion Criteria:

* Initial indication for IFX being predominantly fistulizing perianal disease.
* Any contraindications for continuing IFX treatment, including prior acute or delayed infusion reaction to a TNF- inhibiting agent, any active infection requiring parenteral or oral antibiotic treatment, known infection with tuberculosis, human immunodeficiency virus (HIV) or hepatitis virus.
* Any condition including physician finds incompatible with participation in the study or the patient being unwilling or unable to follow protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Time to relapse after discontinuation of IFX | 48 weeks
  Relapse defined as CDAI >150 and an increase in CDAI from baseline >70 over 2 consecutive weeks (or definitive relapse as judged by treating physician)

SECONDARY OUTCOMES:
Time to loss of remission | 48 weeks
  Loss of remission defined as CDAI > 150
Proportion of patients who maintain clinical remission | 48 weeks
  Defined as CDAI<150
Proportion of patients who maintain clinical and endoscopic remission | 48 weeks
  Defined as CDAI<150 and SES-CD ≤ 2
Proportion of patients who experience relapse (more stringent definition) | 48 weeks
  Relapse defined as CDAI >150 and an increase in CDAI from baseline >100 over 2 consecutive weeks (or definitive relapse as judged by treating physician)
Proportion of patients who experience relapse | 48 weeks
  Relapse defined as CDAI >150 and an increase in CDAI from baseline >70 over 2 consecutive weeks (or definitive relapse as judged by treating physician)drug therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ainsworth, MD.PHD.,DMSc, Principal Investigator — Herlev Hospital, dep. of gastroenterology medical section.
Locations (13):
- Denmark (9):
  - Aarhus University Hospital, Aarhus, Aarhus C
  - Bispebjerg Hospital, Copenhagen, Copenhagen NV
  - Nykøbing F. Sygehus, Nykøbing Falster, Nykøbing
  - Odense University hospital, Odense, Odense C
  - Herlev Hospital, department of gastroenterology medical section, Herlev
  - Hospital enheden vest Herning, Herning
  - Hvidovre Hospital, Hvidovre
  - Silkeborg Regional Hospital, Diagnostic Center, Silkeborg
  - Slagelse Sygehus, Slagelse
- Helsinki University Hospital and University of Helsinki, Helsinki, Finland
- Akerhus University Hospital, Oslo, Norway
- Sweden (2):
  - Skane University Hospital, Lund
  - Karolinska Institute, Stockholm

REFERENCES:
- [Derived] Buhl S, Steenholdt C, Brynskov J, Christensen KR, Dorn-Rasmussen M, Thomsen OO, Bendtzen K, Klausen TW, Dahlerup JF, Thorsgaard N, Jahnsen J, Molazahi A, Pedersen N, Kjeldsen J, Almer S, Dahl EE, Vind I, Cannon AG, Marsal J, Sipponen T, Agnholt JS, Kievit HAL, Aure SL, Martinsen L, Meisner S, Hansen JM, Ainsworth MA. Discontinuation of Infliximab Therapy in Patients with Crohn's Disease. NEJM Evid. 2022 Aug;1(8):EVIDoa2200061. doi: 10.1056/EVIDoa2200061. Epub 2022 Jun 14. PMID 38319804
- [Derived] Buhl SS, Steenholdt C, Brynskov J, Thomsen OO, Bendtzen K, Ainsworth MA. Discontinuation of infliximab therapy in patients with Crohn's disease in sustained complete remission (the STOP IT study): protocol for a double-blind, randomised, placebo-controlled, multicentre trial. BMJ Open. 2014 Dec 18;4(12):e005887. doi: 10.1136/bmjopen-2014-005887. PMID 25524543

DOCUMENTS (2):
  • Study Protocol (2015-10-19): https://cdn.clinicaltrials.gov/large-docs/26/NCT01817426/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/26/NCT01817426/SAP_001.pdf